CLINICAL TRIAL: NCT02581150
Title: Cost-utility Analysis of the Outpatient Hospitalization Versus Conventional Hospitalization in Endovascular Treatment of Occlusive Arterial Disease
Brief Title: Cost-utility Analysis of the Outpatient Versus Conventional Hospitalization in Treatment of Occlusive Arterial Disease
Acronym: AMBUVASC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC15_0044; PRME-14-0444 (Other Grant/Funding Number: French Minstry of Health)
Record Dates: First submitted 2015-10-19; First posted 2015-10-20 (Estimated); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Peripheral Arterial Disease
Keywords: Outpatient hospitalization; Randomized trial; Peripheral arterial disease; Endovascular treatment; Health Economics
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Outpatient hospitalisation (Other): The intervention is the Treatment of Occlusive Arterial Disease, during an ambulatory hospitalisation, with the use of an arterial closure device (ACD).
  The patients treated for PAD (Peripheral Arterial Disease) are informed and prepared in the morning of D0. The surgical endovascular procedure is performed at D0 before 1:00 p.m. The patients leave the hospital in the evening at D0 after a systematic visit.
  Interventions: Procedure: Treatment of Occlusive Arterial Disease
- Conventional inpatient hospitalisation (Other): The intervention is the Treatment of Occlusive Arterial Disease, during a conventional hospitalisation, with or without ACD (ACD will be used at the discretion of the interventionalist).
  The patients treated for PAD arrive at the hospital the day before surgery (D-1). The surgical endovascular procedure takes place the next day (D0). The day after (D1), the patients leave the hospital after a systematic visit.
  Interventions: Procedure: Treatment of Occlusive Arterial Disease

INTERVENTIONS:
Procedure: Treatment of Occlusive Arterial Disease — Regarding the intervention, the technique used during the diagnostic and/or therapeutic procedure shall be left to the operator's discretion, except the use of an arterial closure device (ACD). In the ambulatory hospitalisation arm, the ACD use will be mandatory. In the conventional hospitalisation arm, ACD will be used at the discretion of the interventionalist.

SUMMARY:
The purpose of this study is to assess the efficiency of outpatient surgery compared to conventional hospitalization in endovascular treatment of occlusive arterial disease. A cost-utility analysis will be conducted from a societal perspective. Patients referred for peripheral arterial disease (PAD) will be randomized in two arms and a 3 months follow-up will be performed.

DETAILED DESCRIPTION:
Rationale for ambulatory hospitalization is based on increased demand of hospital care, hospital budgets constraints and patients who ask for a prompt recovery. Consequently, physicians should find ways to optimize the resources' allocation, without compromising quality, safety and efficiency of patient care. Several studies and routine practice have shown that ambulatory hospitalization was safe but we are still lacking evidence to demonstrate the cost-utility of this kind of management.

ELIGIBILITY:
Inclusion Criteria:

* Patients limping
* Patients with PAD requiring endovascular management
* Patients with stabilized level 1 to 3 ASA (classification of the American Society of Anesthesiology)
* Ability to walking
* Endovascular indicated and compatible with an introducer 5F to 7F
* Agreeing to participate in the study and having signed an informed consent.
* Agreeing to lend itself to a post-operative monitoring a duration of 30 days
* Social Insured

Exclusion Criteria:

* No possibility of an outpatient management
* Previous participation in the AMBUVASC study
* Refusal of patient to participate in the study
* Patient with hemostasis disorders
* Acute Ischemia
* Using a more 7F introducer
* Radial or brachial puncture
* Antegrade femoral puncture
* Contraindication to endovascular treatment
* Less than one month life expectancy
* Participation in another clinical trial

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2016-02; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Incremental Cost Effectiveness Ratio (ICER) comparing cost and utility in the two arms | 3 months
  The objective of the study is to perform a cost-utility analysis comparing outpatient surgery to conventional hospitalization in endovascular treatment of occlusive arterial disease. The analysis will be conducted from a society's perspective using a one-month time horizon following the date of intervention (and 2 months before intervention). A microcosting approach will be used to estimate the cost of the surgical intervention in both arms and all subsequent in-hospital and ambulatory care resources consumption will be systematically recorded during the one month follow-up period. Effectiveness will be assessed in terms of Quality-Adjusted Life-Years (QALYs) estimated from patients' answers to the Euroqol EQ-5D questionnaire and french preferences scores. Results will be presented as an incremental cost-per-QALY ratio.

SECONDARY OUTCOMES:
Budget impact analysis | 5 years
  The budget impact analysis will estimate the net financial profit (the difference between the costs incurred and profits obtained, or avoided costs) in developing the ambulatory surgery in the management of PAD. The perspective adopted will be that of the health care facilities and of the National health insurance. This analysis will be conducted in a 5 years time horizon to consider a full exploitation of the potential for substitution between conventional hospitalisation and ambulatory hospitalisation for eligible patients.
Complication rates | 1 month
  The major vascular complications that can occur within 30 days are: Complications Intraoperative, Hematoma, Bleeding from the groin, arteriovenous fistula, Pseudo aneurysm, retroperitoneal hemorrhage, Critical Ischemia, Infection, Thrombosis.
Functional improvement | 1 month
  The assessment of the functional improvement will be performed with Rutherford Classification.
Time period to back-to-work | 1 month
  The time period to back-to-work will be assessed through the measurement of the duration of sick leave for people who work.

CONTACTS AND LOCATIONS:
Overall Officials: Yann Gouëffic, Md., PhD., Principal Investigator — University Hospital of Nantes, France
Locations (11):
- France (11):
  - Besançon University Hospital, Besançon
  - Colmar Hospital, Colmar
  - Dijon University Hospital, Dijon
  - Clinique de Fontaine, Fontaine-lès-Dijon
  - La Roche sur Yon Hospital, La Roche-sur-Yon
  - Marseille University Hospital (La Timone), Marseille
  - Marseille University Hospital (North), Marseille
  - Nantes University Hospital, Nantes
  - Rennes University Hospital, Rennes
  - Rouen Clinique de l'Europe, Rouen
  - Saint-Etienne University Hospital, Saint-Etienne